CLINICAL TRIAL: NCT00070811
Title: Functional Outcomes of Cleft Lip and Lip Revision Surgery
Brief Title: Assessing the Results of Lip Surgery in Patients With Cleft Lip and Palate
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Carroll-ann Trotman, DDS, Adjunct Professor, Department of Orthodontics, University of North Carolina, Chapel Hill
Other Study IDs: NIDCR-13814; R01DE013814 (NIH)
Record Dates: First submitted 2003-10-08; First posted 2003-10-13 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Cleft Lip; Cleft Lip and Palate
Keywords: Facial form; Facial animation; Lip muscle reconstruction; Lip form; Lip function
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Revision: Patients with repaired cleft lip who receive lip revision surgery
  Interventions: Procedure: Lip revision surgery
- Non-Revision: Patients with repaired cleft lip who do not have lip revision surgery
- Non-cleft: Non-cleft 'control' subjects.

INTERVENTIONS:
Procedure: Lip revision surgery — Full or partial muscle thickness lip revision surgery.
  Other Names: Primary lip repair; Secondary lip repair
  Groups: Revision

SUMMARY:
The purpose of this study is to determine whether secondary (revision) surgery to the lip in patients with cleft lip and palate is effective in improving lip function and appearance.

DETAILED DESCRIPTION:
Children born with clefting of the upper lip exhibit obvious disfigurement of the upper lip and nose. As illustrated below, primary lip surgery of the infant dramatically improves the severe deformity of the perioral and nasal region. It is widely recognized, however, that most patients require additional lip surgeries for an optimum esthetic result. Clinicians often disagree as to when this end point is reached since the decision for additional lip revision is based on subjective clinical assessments.

Facial morphology during function has a major impact on how a person is perceived in society and is known to be an important component of the esthetic outcome for cleft patients, but it has been particularly difficult to incorporate measures of lip function into the decision-making process. It is likely that the different surgical procedures for both primary lip closure and secondary lip revision could be improved if the effects of alternative surgical techniques on function were better understood. The subjects for this project consist of two cleft lip and palate patient groups treated at the University of North Carolina (UNC) Craniofacial Center: one cleft group will be patients who are candidates for additional lip revision surgery; the other cleft group will be patients who have been judged not to need lip revision; and a matched non-cleft group who present for routine dental care at UNC School of Dentistry. The goals of this project are to objectively measure and quantify functional facial impairment in cleft patients, and to establish more reliable, functionally relevant outcome criteria for treatment planning and evaluation of these individuals. Our specific aims, therefore, are to

1. In a prospective non-randomized controlled clinical trial, evaluate the efficacy of lip revision surgery by a) Examining longitudinal changes in function after lip revision, and b) Examining whether the change in function after lip revision differs from the change that would be observed due to maturation only in the matched non-cleft 'normal' group, and the change in the cleft but non-lip revised group.
2. a) Estimate the effect of cleft lip and palate on function after primary lip and palate repair but prior to lip revision surgery by comparing those patients scheduled to receive a lip revision with those who are judged not to need a lip revision, and b) Estimate the impairment in function in cleft lip and palate patients without lip revision relative to matched non-cleft subjects.
3. Compare the assessments of dynamic lip function provided by objective measures with subjective clinical judgments/ratings of craniofacial plastic surgeons who perform lip revision surgery, and evaluate the potential of the new methods for clinical application.
4. Evaluate whether objective information when added to the clinician's subjective evaluation of a patient alters the surgical treatment plan or the goals of treatment when subjective and objective information are incorporated in the decision-making and treatment planning process. This specific aim will be useful in adapting and assessing the potential of the new objective methods for application in a clinical setting.
5. To establish 'parameters of care' criteria for secondary lip revision treatment decision-making based on standardized, systematic subjective evaluation, and an objective measurement of movement capacity during function of the upper lip.
6. Assess the long-term effects of maturation on function following lip revision by continuing data-collection beyond the one-year post-revision on patients recruited during the period of the initial grant and long-term follow-up (18 and 30 months) on newly recruited lip revision patients, and in so doing, evaluate the efficacy of cleft lip revision surgery.

To address these aims, we have identified a group of highly qualified individuals with widely recognized expertise in the application of the proposed methodologies, and a panel of surgeons experienced in cleft care for clinical evaluation of outcomes. This expertise, the availability of an appropriate patient resource, and the home institution's 40-year history of strong commitment to the care of these patients and craniofacial research, all favor success in meeting the goals of the project.

ELIGIBILITY:
1. Children:

   Cleft lip and palate revision and non-revision patients.

   Inclusion criteria:
   * A previously-repaired complete unilateral or bilateral cleft lip and cleft palate;
   * For the lip revision patients, the professional clinical recommendation by the Center's craniofacial plastic surgeon for a full-thickness lip revision;
   * Patient interest / parent willingness to participate in the study;
   * An ability to comprehend verbal instructions; and
   * An age range of 5-17 yrs.

   Exclusion criteria:
   * The presence of an isolated cleft lip;
   * Previous lip-revision surgery or other facial soft-tissue surgery;
   * Previous orthognathic surgery;
   * A diagnosis of a craniofacial anomaly other than cleft lip and palate;
   * A medical history of diabetes, collagen vascular disease, systemic neurologic impairment; or
   * Mental or hearing impairment to the extent that comprehension or ability to perform the tests is hampered.

   Non-cleft subjects.

   Inclusion criteria:
   * Patient interest / parent willingness to participate in the study;
   * An ability to comprehend verbal instructions; and
   * An age range of 5-17 yrs.

   Exclusion criteria:
   * Previous orthognathic or facial soft-tissue surgery;
   * A medical history of diabetes, collagen vascular disease, systemic neurologic impairment; or
   * Mental or hearing impairment to the extent that comprehension or ability to perform the tests is hampered.
2. Infants

Cleft lip and palate patients.

Inclusion Criteria:

* The professional clinical recommendation by the Center's craniofacial plastic surgeon for a cleft lip repair surgery;
* Parent willingness to have baby participate in the study;
* An age range of 0-6 months.

Exclusion Criteria:

* Has had surgery for any reason
* A diagnosis of a craniofacial anomaly other than cleft lip and palate;
* A medical history of diabetes, collagen vascular disease, and systemic neurologic impairment

Non-cleft subjects.

Inclusion Criteria:

* Parent willingness to have baby participate in the study;
* An age range of 0-6 months.

Exclusion Criteria

* Has had surgery for any reason including bone surgery
* A medical history of diabetes, collagen vascular disease, and systemic neurological impairment

Ages: 3 Months to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects will be recruited and screened mainly in the UNC Craniofacial Center, the Graduate Orthodontic Clinic, the Pediatric Dentistry Clinic, and the Orthodontic Faculty Practice of the University of North Carolina.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2001-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Facial movement/animation | 6

SECONDARY OUTCOMES:
Lip Force | 6
EMG | 6
Lip sensation | 6

CONTACTS AND LOCATIONS:
Overall Officials: Carroll-Ann Trotman, BDS, MA, MS, Principal Investigator — University of NC at Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Andreatta RD, Barlow SM. Somatosensory gating is dependent on the rate of force recruitment in the human orofacial system. J Speech Lang Hear Res. 2009 Dec;52(6):1566-78. doi: 10.1044/1092-4388(2009/08-0116). Epub 2009 Aug 28. PMID 19717653
- [Background] Trotman CA, Faraway JJ, Essick GK. Three-dimensional nasolabial displacement during movement in repaired cleft lip and palate patients. Plast Reconstr Surg. 2000 Apr;105(4):1273-83. doi: 10.1097/00006534-200004040-00003. PMID 10744215
- [Background] Trotman CA, Faraway JJ, Silvester KT, Greenlee GM, Johnston LE Jr. Sensitivity of a method for the analysis of facial mobility. I. Vector of displacement. Cleft Palate Craniofac J. 1998 Mar;35(2):132-41. doi: 10.1597/1545-1569_1998_035_0132_soamft_2.3.co_2. PMID 9527310
- [Background] Trotman CA, Faraway JJ. Sensitivity of a method for the analysis of facial mobility. II. Interlandmark separation. Cleft Palate Craniofac J. 1998 Mar;35(2):142-53. doi: 10.1597/1545-1569_1998_035_0142_soamft_2.3.co_2. PMID 9527311
- [Background] Liu J, Xu HH, Zhou H, Weir MD, Chen Q, Trotman CA. Human umbilical cord stem cell encapsulation in novel macroporous and injectable fibrin for muscle tissue engineering. Acta Biomater. 2013 Jan;9(1):4688-97. doi: 10.1016/j.actbio.2012.08.009. Epub 2012 Aug 16. PMID 22902812
- [Background] Liu J, Zhou H, Weir MD, Xu HH, Chen Q, Trotman CA. Fast-degradable microbeads encapsulating human umbilical cord stem cells in alginate for muscle tissue engineering. Tissue Eng Part A. 2012 Nov;18(21-22):2303-14. doi: 10.1089/ten.TEA.2011.0658. Epub 2012 Jul 19. PMID 22697426
- [Result] Trotman CA, Phillips C, Essick GK, Faraway JJ, Barlow SM, Losken HW, van Aalst J, Rogers L. Functional outcomes of cleft lip surgery. Part I: Study design and surgeon ratings of lip disability and need for lip revision. Cleft Palate Craniofac J. 2007 Nov;44(6):598-606. doi: 10.1597/06-124.1. PMID 18177192
- [Result] Trotman CA, Faraway JJ, Losken HW, van Aalst JA. Functional outcomes of cleft lip surgery. Part II: Quantification of nasolabial movement. Cleft Palate Craniofac J. 2007 Nov;44(6):607-16. doi: 10.1597/06-125.1. PMID 18177193
- [Result] Essick GK, Phillips C, Trotman CA. Functional outcomes of cleft lip surgery. Part IV: Between- and within-participant variables affecting lip vermilion sensory thresholds. Cleft Palate Craniofac J. 2007 Nov;44(6):624-34. doi: 10.1597/06-129.1. PMID 18177194
- [Result] Trotman CA, Barlow SM, Faraway JJ. Functional outcomes of cleft lip surgery. Part III: Measurement of lip forces. Cleft Palate Craniofac J. 2007 Nov;44(6):617-23. doi: 10.1597/06-138.1. PMID 18177195
- [Result] Trotman CA, Faraway JJ, Phillips C. Visual and statistical modeling of facial movement in patients with cleft lip and palate. Cleft Palate Craniofac J. 2005 May;42(3):245-54. doi: 10.1597/04-010.1. PMID 15865457
- [Result] Essick GK, Dorion C, Rumley S, Rogers L, Young M, Trotman CA. Report of altered sensation in patients with cleft lip. Cleft Palate Craniofac J. 2005 Mar;42(2):178-84. doi: 10.1597/03-124.1. PMID 15748109
- [Result] Trotman CA, Phillips C, Faraway JJ, Ritter K. Association between subjective and objective measures of lip form and function: an exploratory analysis. Cleft Palate Craniofac J. 2003 May;40(3):241-8. doi: 10.1597/1545-1569_2003_040_0241_absaom_2.0.co_2. PMID 12733951
- [Result] Ritter K, Trotman CA, Phillips C. Validity of subjective evaluations for the assessment of lip scarring and impairment. Cleft Palate Craniofac J. 2002 Nov;39(6):587-96. doi: 10.1597/1545-1569_2002_039_0587_voseft_2.0.co_2. PMID 12401105
- [Result] Lee JY, Han Q, Trotman CA. Three-dimensional facial imaging: accuracy and considerations for clinical applications in orthodontics. Angle Orthod. 2004 Oct;74(5):587-93. doi: 10.1043/0003-3219(2004)0742.0.CO;2. PMID 15529491
- [Result] Faraway JJ, Trotman CA. Shape change along geodesics with application to cleft lip surgery. J R Stat Soc Ser C Appl Stat. 2011 Nov;60(5):743-755. doi: 10.1111/j.1467-9876.2011.01017.x. Epub 2011 Sep 29. PMID 22639469
- [Result] Trotman CA. Faces in 4 dimensions: Why do we care, and why the fourth dimension? Am J Orthod Dentofacial Orthop. 2011 Dec;140(6):895-9. doi: 10.1016/j.ajodo.2011.07.014. PMID 22133956
- [Result] Barlow SM, Trotman CA, Chu SY, Lee J. Modification of perioral stiffness in patients with repaired cleft lip and palate. Cleft Palate Craniofac J. 2012 Sep;49(5):524-9. doi: 10.1597/10-092. Epub 2011 Jan 19. PMID 21247345
- [Result] Tanikawa C, Takada K, van Aalst J, Trotman CA. Objective three-dimensional assessment of lip form in patients with repaired cleft lip. Cleft Palate Craniofac J. 2010 Nov;47(6):611-22. doi: 10.1597/09-099. Epub 2010 Mar 12. PMID 20500076
- [Result] Trotman CA, Faraway JJ, Phillips C, van Aalst J. Effects of lip revision surgery in cleft lip/palate patients. J Dent Res. 2010 Jul;89(7):728-32. doi: 10.1177/0022034510365485. Epub 2010 May 3. PMID 20439935
- [Result] Chu SY, Barlow SM, Lee J. Nonparticipatory stiffness in the male perioral complex. J Speech Lang Hear Res. 2009 Oct;52(5):1353-9. doi: 10.1044/1092-4388(2009/08-0101). Epub 2009 Aug 28. PMID 19717655
- [Result] Weismer G, Barlow S, Smith A, Caviness J. Special Panel Session: Driving Critical Initiatives in Motor Speech. J Med Speech Lang Pathol. 2008;16(4):283. PMID 19421339
- [Result] Chu SY, Barlow SM, Kieweg D, Lee J. OroSTIFF: Face-referenced measurement of perioral stiffness in health and disease. J Biomech. 2010 May 28;43(8):1476-82. doi: 10.1016/j.jbiomech.2010.01.037. Epub 2010 Feb 24. PMID 20185131
- [Result] Essick G, Phillips C, Chung Y, Trotman CA. Effects of lip revision surgery on long-term orosensory function in patients with cleft lip/palate. Cleft Palate Craniofac J. 2013 Sep;50(5):507-12. doi: 10.1597/11-247. Epub 2012 Aug 20. PMID 22906391
- [Result] Trotman CA, Faraway J, Soltmann R, Hartman T, van Aalst J. Facial soft tissue dynamics before and after primary lip repair. Cleft Palate Craniofac J. 2013 May;50(3):315-22. doi: 10.1597/12-080. Epub 2012 Oct 10. PMID 23050657